CLINICAL TRIAL: NCT03476993
Title: Open-label Non-comparative Study to Evaluate the Efficacy and Safety of BCD-085 (JSC BIOCAD, Russia) in Combination With Ursodeoxycholic Acid in Patients With Primary Biliary Cholangitis
Brief Title: Non-comparative Study of BCD-085 in Combination With UDCA in Patients With Primary Biliary Cholangitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponosor's decision
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-085-6
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: primary biliary cholangitis; IL-17 monoclonal antibody
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD-085 (Experimental): All patients will receive BCD-085 (subcutaneous injection) in combination with ursodeoxycholic acid (UDCA) in standard dose 13-15 mg/kg/day
  Interventions: Biological: BCD-085

INTERVENTIONS:
Biological: BCD-085 — All patients will receive BCD-085 (subcutaneous injections) once a week during the period of induction of remission, then once every 2 weeks during the period of remission maintenance and then once every 4 weeks during the period of accumulation of treatment effect. All patients will receive ursodeoxycholic acid (UDCA) in standard dose 13-15 mg/kg/day.

SUMMARY:
BCD-085 is an innovative drug, anti-interleukin-17 monoclonal antibody. The aim of the study is to evaluate the efficacy and safety of BCD-085 in patients with primary biliary cholangitis (PBC).

DETAILED DESCRIPTION:
This is an open-label proof-of-concept phase 2A study. The aim of the study is to evaluate the efficacy and safety of BCD-085 in combination with ursodeoxycholic acid in patients with primary biliary cholangitis (PBC) with compensated liver function with an inadequate (suboptimal) response to ursodeoxycholic acid.

In this study the inadequate (suboptimal) response to ursodeoxycholic acid (UDCA) is defined as screening alkaline phosphatase (ALP) level > 1.67 ULN (the upper limit of normal) despite treatment with UDCA in stable dose for at least 6 months before signing the ICF.

ELIGIBILITY:
Inclusion Criteria:

1. Singed informed consent form (ICF)
2. Men and women, age 18 - 80 years at the time of signing the ICF
3. Established diagnosis of PBC with following criteria (according to EASL 2017 guidelines):

   * documented ALP elevation
   * documented АМА ≥ 1:40 or PBC-specific ANА (anti-sp100/anti-gp210).
4. Suboptimal response to ursodeoxycholic acid (UDCA) taken in stable dose for at least 6 months before signing ICF with screening alkaline phosphatase (ALP) level > 1.67 ULN (the upper limit of normal)
5. Fertile patients and their partners agree to use barrier contraception throughout the study and 4 weeks after its completion.

Exclusion Criteria:

1. History of gastrointestinal bleeding, hepatic encephalopathy or ascites requiring treatment with diuretics.
2. MELD ≥ 15, history of liver transplantation, staying in the Liver Transplant Waiting List.
3. Established diagnosis of hepatocellular carcinoma (HCC), hepatorenal syndrome.
4. Direct bilirubin > 1.0 mg/dL at screening.
5. Documented diagnosis: nonalcoholic steatohepatitis, autoimmune hepatitis, primary sclerosing cholangitis, alcoholic liver disease, Gilbert's syndrome, Wilson disease, hemochromatosis, alfa-1-antitrypsin deficiency.
6. HIV, hepatitis B, hepatitis C or syphilis.
7. Use of colchicine, methotrexate, azathioprine or systemic corticosteroids within 3 months before signing the ICF.
8. Previous use of monoclonal antibodies targeting IL17 or its receptor.
9. Vaccination with live or attenuated vaccines within 8 weeks before signing the ICF.
10. Any active systemic infection or recurrent infection at screening or 30 days before signing the ICF.
11. Established diagnosis of chronic disease (e.g. sepsis, invasive mycosis, histoplasmosis etc.) that may increase the risk of infectious adverse events during the study.
12. Severe infections (including those that required hospitalization or parenteral antibacterial/antimycotic/antiprotozoal treatment) within 6 months before signing the ICF
13. Established diagnosis of herpes zoster infection (or history of herpes zoster infection).
14. latent tuberculosis infection (positive results of the Diaskintest or QuantiFERON test, or T-spot).
15. Concurrent diseases at screening that may increase the risk of adverse events during the study or affect the evaluation of PBC symptoms (mask, enhance or alter the symptoms of PBC, or cause clinical or laboratory signs/symptoms similar to those of PBC)
16. Known allergy or intolerance to monoclonal antibody drugs (murine, chimeric, humanized, or human) or any other components of BCD-085.
17. Pregnancy, breastfeeding or planning of pregnancy during the study.
18. Any psychiatric conditions including severe depressive disorders and/or any history of suicidal thoughts or suicidal attempts that may constitute the excessive risk for the patient or that may affect the patient's ability to follow the protocol.
19. Alcohol or substance abuse.
20. Participation in other clinical trials within less than 90 days before signing the ICF.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with alkaline phosphatase (ALP) decrease > 40% from Baseline (day 1 week 0) or with normal ALP level (Barcelona criteria) after 24 weeks of treatment with BCD-085 in combination with UDCA. | week 24
  Biochemical response is defined as ALP decrease > 40% from Baseline or normalisation of ALP level (Barcelona criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Marina Maevskaya, Principal Investigator — State Budgetary Higher Vocational Education Institution I.M. Sechenov First Moscow State Medical University
Locations (3):
- Russia (3):
  - State Budgetary Higher Vocational Education Institution I.M. Sechenov First Moscow State Medical University, Moscow
  - North-Western State Medical University named after I.I. Mechnikov, Saint Petersburg
  - Smolensk state medical university, Smolensk

IPD SHARING:
Plan to Share IPD: No